CLINICAL TRIAL: NCT03959813
Title: Evaluation of the Impact of Psychomotricity on the Patients Body Experience in Palliative Care
Acronym: PSYCHOMOTPAL
Status: Withdrawn | Type: Observational
Why Stopped: the ethics committee has not accepted the extension
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7254
Record Dates: First submitted 2019-05-06; First posted 2019-05-22 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Palliative Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Psychomotricity by touching and passive mobilizations — The patient will have a first psychomotricity session. It will be carried out remotely from the drug catches to avoid bias induced by their administration having effects on the symptoms studied.
  Before and after the session, two evaluations will be offered to the patient and performed by a nurse:
  * A questionnaire, based on the physical experience,
  * The ESAS scale will be administered to the patient to assess the importance of symptoms (pain, depression, anxiety, discomfort) During the session, a touch treatment will be offered to promote awareness of the body. Passive mobilizations at the level of the members and the axis will then be proposed, to promote the pleasure of being in motion. A touch treatment will be done again to promote relaxation.
  A questionnaire can be offered to the patient after 4 sessions to assess his perception of psychomotricity.

SUMMARY:
Palliative care is part of a comprehensive approach to the person, in the advanced phase of a serious illness. The purpose of this care is to relieve painful symptoms, to promote comfort and quality of life. In the context of a serious illness, the sick person is confronted with body modifications that have an impact on his body experience, that is, on his feelings and on the image that he has of his body.

Psychomotricity is a paramedical discipline that focuses on body-psyche links. The psychomotor therapist is authorized to take care of psychomotor disorders, as defined in the decree of competences. These psychomotor disorders appear in connection with the evolution of the serious illness and the presence of symptoms in these patients (ex: disorders of the tonic regulation, psychomotor disharmony, disorders of the representation of the body, etc.). In palliative care, the psychomotor therapist seeks to regulate these psychomotor disorders and thus to promote a more satisfying physical experience in the patient, through the use of different bodily approaches.

Several studies have shown the beneficial effects of touching and moving the body in cancer patients, but no work evaluating the effects of the psychomotor approach (involving various body mediations) on the body experience of patients with cancer in palliative situation

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Man or woman
* Subject who has agreed to participate in the research and to use the data collected for research purposes
* Patient with solid cancer or hematological malignancy in palliative stage, that is to say a cancerous disease for which no curative treatment is no longer envisaged, with committed vital prognosis
* Hospitalize patient in palliative care unit
* Patient with indication of care in psychomotricity defined by the decree of competence Decree n ° 88-659 of May 6, 1988
* Patient with a minimum score of 4 on an item or a minimum score of 4 on several cumulative items (with a minimum of 2 on at least one of the items), on the ESAS scale, among the following themes: pain, anxiety, depression, uneasy feeling

Exclusion Criteria:

* Patient whose clinical condition (left to the decision of the investigator) does not allow to perform a psychomotor care and / or participate in a recorded interview (extreme fatigue, confusion, painful uncontrolled symptoms)
* Communication difficulties, patient not speaking or not understanding French
* Impossibility of giving the patient informed information (subject in emergency situation, difficulties in understanding the subject, etc.)
* Patient under guardianship, curatorship
* Patient not affiliated to social welfare regime

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients hospitalized in palliative care units
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Realization of a questionnaire, based on the patient's global and physical feeling | 30 minutes before psychomotor care
  questionnaire used to assess the impact of psychomotor care on the body experience of patients with advanced palliative care cancer, in both a physical and psychological dimension
Realization of a questionnaire, based on the patient's global and physical feeling | 30 minutes after psychomotor care
  questionnaire used to assess the impact of psychomotor care on the body experience of patients with advanced palliative care cancer, in both a physical and psychological dimension

IPD SHARING:
Plan to Share IPD: No